CLINICAL TRIAL: NCT04922164
Title: Using Cueing Interventions to Bridge Intention-behaviour Gaps: an Longitudinal Experimental Study on Promoting Breastfeeding
Brief Title: Using Cueing Interventions to Promote Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Qiuyan Liao, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20190320bf
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Receive education-based messages about the health benefit of breastfeeding
- Social normative cues (Other): Receive social normative cues related to breastfeeding
  Interventions: Behavioral: Cue intervention
- Goal-related cues (Other): Receive goal-related cues related to breastfeeding
  Interventions: Behavioral: Cue intervention

INTERVENTIONS:
Behavioral: Cue intervention — Around 30 pieces of narrative information about how a mother behaves in specific decision context will be derived from our qualitative study to construct social normative cues.
  For goal-related cues, words relating to each category of breastfeeding-related values, benefits and goals will be identified and used to construct the messages (e.g. "attractive body shape", "smart baby", "natural", "strong immunity" and etc.). Each goal-priming message will be presented with brief priming words and a picture of an image of the desirable goal.
  Arms: Goal-related cues; Social normative cues

SUMMARY:
Background: Interventions focusing on promoting good behavioural intentions were found to only have small-to-moderate effect sizes on changing the actual behaviours. Self-regulation plays an important role to maintain individual attentions to the distant benefits of healthy behaviours and resist to proximal tempting cues from unhealthy behaviours, and thereby facilitate the translation of good intention into actual behaviours. However, self-regulation resources are limited and can be depleted in certain contexts. Providing environmental cues relevant to the desirable behaviours can activate the nonconscious process and lead to behavioural change without conscious awareness, the underlying mechanism of cueing interventions.

Aims: To test the effectiveness of using two types of cues, social normative and goal-related cues, to activate the nonconscious process for facilitating the translation of intentions into actual behaviours. We hypothesize that (1) cueing interventions will be more effective than will conventional education-based interventions (providing factual information about health benefits) be for changing behaviours; (2) cueing interventions are more effective for participants who have a tendency to use an intuitive mode in information processing; and (3) goal priming is more effective for participants with stronger motivation to pursue the goal of sustaining breastfeeding.

Subject and study design: The hypotheses will be tested in the behavioural context of breastfeeding among first-time mothers because: first, primiparous women may have less self-regulation resources due to high cognitive demand for postpartum adjustment during motherhood transition; and second, while breastfeeding intention and initiation were high, maintaining breastfeeding for the first six months postpartum was generally low in Hong Kong, indicating a substantial intention-behaviour gap. We propose to recruit 600 primiparous women. Baseline assessments will be conducted face-to-face using a standardized questionnaire. Participants will be randomly allocated to the control group (receive education-based messages about the health benefit of breastfeeding) or one of the two intervention groups (receive either social normative cues or goal-related cues related to breastfeeding). All messages will be delivered through smartphone on a daily basis over 16 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* being ≥18 years
* being Chinese ethnicity and Hong Kong residents
* without any serious medical or obstetric complications
* having a full-term (i.e. gestational age ≥37 weeks) healthy infant with normal birthweight (≥2,500 grams)

Exclusion Criteria:

* with linguistic and cognitive barriers impeding completion of face-to-face and telephone interviews or comprehension of the intervention materials
* physical anomalies that contraindicate breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — First-time mothers from the postnatal wards
Enrollment: 252 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
The effectiveness of two cueing interventions, cueing with social norms and goal priming at one month postpartum | Immediately after participants complete the questionnaire
  The name of measurement: exclusive and any breastfeeding duration at one month postpartum
  Unit of measurement: the duration of breastfeeding
The effectiveness of two cueing interventions, cueing with social norms and goal priming at three months postpartum | Immediately after participants complete the questionnaire
  The name of measurement: exclusive and any breastfeeding duration at three months postpartum
  Unit of measurement: the duration of breastfeeding
The effectiveness of two cueing interventions, cueing with social norms and goal priming at six months postpartum | Immediately after participants complete the questionnaire
  The name of measurement: exclusive and any breastfeeding duration at six months postpartum
  Unit of measurement: the duration of breastfeeding

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong School of Public Health, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.